CLINICAL TRIAL: NCT07222631
Title: An Open-Label, First-in-Human Phase 1/2, Dose-Escalation and Dose-Expansion/ Combination Therapy Study to Investigate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of SB-4826 as a Single Agent in Adult Participants With Locally Advanced or Metastatic Solid Tumors or Non-Hodgkin Lymphomas and in Combination With Rituximab in Adult Participants With Non-Hodgkin Lymphomas.
Brief Title: SB-4826 in Adult Participants With Locally Advanced or Metastatic Solid Tumors or Non-Hodgkin Lymphomas
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: The Institute for Follicular Lymphoma Innovation (Unknown)
Responsible Party: Principal Investigator, Peter Vu, Associate Professor of Medicine, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 812350
Record Dates: First submitted 2025-10-28; First posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Non Hodgkin Lymphoma; Solid Tumor
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Locally advanced or metastatic solid tumors Phase 1 monotherapy (Experimental): Phase 1 dose escalation SB-4826 monotherapy
  Interventions: Drug: SB-4826
- Non-Hodgkin lymphoma Phase 1 monotherapy (Experimental): Phase 1 dose escalation SB-4826 monotherapy
  Interventions: Drug: SB-4826
- Non-Hodgkin lymphoma Phase 1 combination therapy (Experimental): Phase 1 dose escalation SB-4826 in combination with rituximab
  Interventions: Drug: SB-4826; Drug: Rituximab
- Non-Hodgkin lymphoma Phase 2 combination therapy (Experimental): Phase 2 dose expansion SB-4826 in combination with rituximab
  Interventions: Drug: SB-4826; Drug: Rituximab

INTERVENTIONS:
Drug: SB-4826 — Small ubiquitin-like modifier E1 inhibitor
Drug: Rituximab — Cluster of differentiation 20 blocker
  Other Names: Rituxan
  Arms: Non-Hodgkin lymphoma Phase 1 combination therapy; Non-Hodgkin lymphoma Phase 2 combination therapy

SUMMARY:
The goal of this clinical trial is to learn what dose of the drug SB-4826 can be given safely in patients with solid tumors and non-Hodgkin lymphomas. This drug will be used alone in patients with solid tumors, and will be used alone or in combination with rituximab in patients with non-Hodgkin lymphomas. The main questions this clinical trial aims to answer are:

What is the maximum dose of SB-4826 that can be used safely in patients with solid tumors and non-Hodgkin lymphomas, and will it work? How does SB-4826 work in people with cancer? How is SB-4826 absorbed, broken down, and excreted by the body?

Participants will:

Take drug SB-4826 every other day for up to 1 year; keep a diary of when they take SB-4826 at home; visit the clinic for checkups, tests, and fill out study questionnaires.

DETAILED DESCRIPTION:
This is a first-in-human, phase 1/2, dose-escalation and dose-expansion / combination therapy study designed to investigate the safety, tolerability, pharmacokinetics, pharmacodynamics, and efficacy of the first-in-class orally bioavailable small ubiquitin-like modifier (SUMO) E1 inhibitor SB-4826, alone and in combination with rituximab (or biosimilar). SUMO E1 inhibitors are a class of anticancer therapies that activate anti-tumor immunity and can directly inhibit the proliferation and survival of cancer cells. SB-4826 is the first SUMO E1 inhibitor that acts through a covalent, allosteric, mechanism.

Phase 1 (Dose-Escalation)

Dose-escalation will include participants with locally advanced or metastatic solid tumors (other than tumors of the brain or central nervous system) or non-Hodgkin lymphoma. Participants with solid tumors will receive only SB-4826 monotherapy, while participants with non-Hodgkin lymphoma will receive either SB-4826 monotherapy or SB-4826 in combination with rituximab.

Participants in the monotherapy treatment group will receive one of an anticipated seven dose-levels ranging from 20 to 600 mg SB-4826 twice weekly. The seven dose-escalation levels include: 20, 40, 80, 140, 240, 400, and up to 600 mg. The selection of the dose-level above 400 mg will be based on the review of the cumulative safety (through the dose-limiting toxicity period) and available pharmacokinetic and pharmacodynamic data from the previous treatment groups.

The recommended phase 2 dose will be the optimal biological dose as determined by the sponsor/principal investigator (based on recommendation from the safety review committee) and consideration of all safety information (e.g., dose limiting toxicity, maximum tolerated dose, treatment-related adverse events) together with available pharmacokinetic, pharmacodynamic, and efficacy data. The recommended phase 2/optimal biological dose may be the maximum tolerated dose or may be a lower dose where optimal pharmacodynamic and pathway inhibition are observed. The recommended phase 2 dose will not exceed the maximum tolerated dose.

Enrollment in the combination group will start after the recommended phase 2 dose is determined for the monotherapy group.

Participants with non-Hodgkin lymphoma in the combination therapy group will receive one of up to 3 dose-levels of SB-4826 twice a week (beginning one dose-level below the monotherapy recommended phase 2 dose) plus rituximab. The recommended phase 2 dose for combination therapy will be determined independently and may be the same or different than the recommended phase 2 dose for monotherapy.

In both phases, dose escalation will be based on a Bayesian Optimal Interval design with a target toxicity rate of 30%. The dose-escalation design will begin with SB-4826 as a single agent (monotherapy). Dose-escalation begins with a single participant enrolled at the first dose-level then proceeds to another single participant enrolled at the next dose-level until dose level 3 (80 mg) is reached or a Grade ≥ 2 adverse event is observed, regardless of attribution, at which time the cohort size switches to 3, and 2 additional participants are added at this dose level to complete the cohort of 3. Once the cohort size is increased to 3, dose escalation and de-escalation decisions are made as follows: If the observed dose limiting toxicity rate at the current dose is less than 23.6% then escalate; if the observed dose limiting toxicity rate at the current dose is greater than 35.8% then de-escalate; and if the observed dose limiting toxicity rate at the current dose is between 23.6% and 35.8%, then add new participants at the current dose. The process ends when either the maximum sample size of 21 has been reached or the sample size at the current dose level reaches the maximum of 12 and the dose limiting toxicity rate at this dose level is between 23.6% and 35.8%. Dose escalation in the combination cohort will proceed similarly, except that the initial cohort size is 3, and the maximum sample size is 9. The maximum tolerated dose is the dose-level determined by the Bayesian Optimal Interval design with a target toxicity rate of 30% within the first 21 days.

Guided by the Bayesian Optimal Interval algorithm, the safety review committee, represented by the UCSD Moores Cancer Center Data and Safety Monitoring Committee, will make recommendations to the sponsor/principal investigator to proceed to the next dose-level or de-escalate to a previous dose-level. Additional responsibilities include making recommendations to add intermediate dose-levels, to add up to 6 additional participants at the anticipated recommended phase 2 dose/optimal biological dose prior to phase 2, to continue or suspend enrollment pending additional information, and making recommendations on defining the recommended phase 2 dose to be used in Phase 2 (Dose-Expansion/ Combination Therapy). Final decisions will be made by the sponsor/principal investigator.

Dose limiting toxicities are pre-defined treatment-related adverse events occurring from first dose of study therapy up to and including Day 21.

Treatment duration will be up to 1 year or until the participant exhibits disease progression, unacceptable toxicity, or other predefined discontinuation or withdrawal criteria are met, whichever occurs first.

Phase 2 (Dose-Expansion/ Combination Therapy)

Phase 2 will enroll only participants with non-Hodgkin lymphomas. They will receive SB-4826 twice a week at the recommended phase 2 dose found in phase 1, in combination with rituximab. Rituximab will be dosed at 375 mg/m^2 intravenously weekly for the first cycle, and then at 375 mg/m^2 intravenously on day 1 starting on cycle 2 for 6 cycles. After 6 cycles, responding participants will transition to maintenance rituximab every 9 weeks for up to 1 year.

Treatment duration will be up to 1 year or until the participant exhibits disease progression, unacceptable toxicity, or other predefined discontinuation or withdrawal criteria are met, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1 - Aged 18 and older.

2- Capable of giving signed informed consent.

3- Phase 1 (Dose-Escalation): Histologically or cytologically confirmed locally advanced or metastatic solid tumor or non-Hodgkin lymphomas. For indolent non-Hodgkin lymphomas, there must be an indication for systemic therapy such as: Local symptoms due to progressive or bulky nodal disease; Threat of or present compromise of normal organ function due to progressive or bulky disease; Presence of systemic B symptoms (ie, fevers, weight loss, night sweats); Presence of symptomatic extranodal disease, such as effusions; Cytopenias due to bone marrow infiltration, autoimmune hemolytic anemia or thrombocytopenia, or hypersplenism; An increase in disease tempo.

4- Phase 2 (Dose-Expansion/ Combination Therapy): Histologically or cytologically confirmed non-Hodgkin lymphomas. For indolent non-Hodgkin lymphomas, there must be an indication for systemic therapy such as: Local symptoms due to progressive or bulky nodal disease; Threat of or present compromise of normal organ function due to progressive or bulky disease; Presence of systemic B symptoms (ie, fevers, weight loss, night sweats); Presence of symptomatic extranodal disease, such as effusions; Cytopenias due to bone marrow infiltration, autoimmune hemolytic anemia or thrombocytopenia, or hypersplenism; An increase in disease tempo. Patients must be planned to receive rituximab as standard of care (on label or medically accepted) treatment for NHL.

5- Participant's malignancy has relapsed after, progressed on, is not a candidate for, is intolerant of, or refuses standard of care therapies.

6- For solid cancer, at least one measurable lesion based on response evaluation criteria in solid tumors (RECIST v1.1).

7- Adequate hematologic parameters unless cytopenia are due to malignancy (i.e. marrow involvement): Hemoglobin ≥ 8 g/dL; Absolute neutrophil count ≥ 1000/microliter or ≥ 750/microliter if Duffy null phenotype; Platelet count ≥ 50,000/microliter.

8- Adequate organ function defined as: Calculated creatinine clearance ≥ 60 mL/min; Serum alanine aminotransferase and aspartate aminotransferase ≤ 1.5 x upper limit of normal; Total bilirubin ≤ 1.5 x upper limit of normal (for participants with known Gilbert's syndrome, direct bilirubin must be ≤ 1.5 x upper limit of normal).

9- All adverse events related to prior therapy or disease (except alopecia) have resolved to grade 2 or less.

10- Life expectancy ≥ 3 months.

11- Eastern Cooperative Oncology Group Performance Status: ≤ 2

12- Female Participants: A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies: Is a woman of nonchildbearing potential (WONCBP) OR is a woman of childbearing potential (WOCBP) and using a contraceptive method that is highly effective (with a failure rate of <1% per year), with low user dependency during the study intervention period and for at least 1 month in the monotherapy group and 12 months in the SB-4826 plus rituximab group. The 1-month timeframe after the last study dose of SB-4826 is a conservative time frame based on the fact that 1 week corresponds to 7 half-lives. Contraception after the last dose of rituximab is required for at least 12 months. The investigator should evaluate the potential for contraceptive method failure (e.g., nonadherence, recently initiated) in relationship to the first dose of study intervention. A WOCBP must have a negative highly sensitive pregnancy test (urine or serum with sensitivity of at least 25 mIU/mL) within 24 hours before the first dose of study drug.

13- Male Participants: Male participants are eligible to participate if they agree to the following during the study intervention period and for at least 3 months after the last study dose. The 3-month timeframe is based on spermatogenesis (74 days) plus at least 1week after the last study dose of SB-4826 (1 week is approximately 7 half-lives). No precautions are required for rituximab. Male participants must refrain from donating sperm plus either be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR agree to use a male condom when having sexual intercourse with a woman of childbearing potential. Female partners of male participants who are WOCBP are permitted to use hormonal contraception and must have barrier method of contraception. Note: A male participant is considered able to father a child unless he has had a bilateral vasectomy with documented aspermia or a bilateral orchiectomy.

Exclusion Criteria:

1. Inability to take oral medications.
2. Use of systemic cancer therapy (e.g., chemotherapy, immunotherapy, biologic, hormonal therapy) within 21 days or 5 half-lives, whichever is shorter.
3. Palliative radiation within 7 days before first dose of study drug.
4. Use of cellular therapy within 60 days before first dose of study drug.
5. Major surgery within 30 days before first dose of study drug.
6. Prior solid organ transplant.
7. Clinically significant cardiovascular disease including any of the following within 6 months before first dose of study drug: myocardial infarction or coronary artery bypass grafting, unstable angina pectoris, serious cardiac ventricular arrhythmia requiring medication, congestive heart failure per New York Heart Association class III or IV, cerebrovascular accident, or poorly controlled hypertension.
8. History of any other malignancy in the past 2 years other than completely resected nonmelanoma skin cancer or carcinoma in situ of the uterine cervix, anus, prostate, bladder, breast, or indolent malignancies that do not require treatment.
9. History of or current chronic liver disease, such as active viral hepatitis, drug- or alcohol-related liver disease, metabolic dysfunction-associated steatohepatitis, autoimmune hepatitis, hemochromatosis, Wilson's disease, alpha-1 antitrypsin deficiency, primary biliary cholangitis, primary sclerosing cholangitis, or any other liver disease considered clinically significant by the investigator.
10. Mean resting corrected QT interval using Fridericia's formula > 470 msec.
11. Active infection that necessitates treatment within 14 days of first dose of study drug.
12. Active hepatitis B or hepatitis C infection regardless of viremia.
13. Known history of human immunodeficiency virus infection with viral load >50 copies/ml at the time of screening.
14. Active autoimmune disease requiring >10 mg of prednisone daily or equivalent, disease-modifying antirheumatic drugs, or immunosuppression.
15. Use of medications that are known to be sensitive narrow therapeutic index or moderate sensitive substrates, strong or moderate inhibitors or strong or moderate inducers of cytochrome P450 3A4/5, or sensitive substrates or inhibitors of P-glycoprotein, breast cancer resistant protein, or organic anion-transporting polypeptide 1B1/1B3 within 14 days or 5 half-lives, whichever is longer, before first dose of study drug.
16. Receipt of any live vaccine (e.g., varicella, pneumococcus) within 30 days of first dose of study drug.
17. Receipt of investigational products, including drugs and devices, within 21 days or five half-lives, whichever is shorter, before first dose of study drug.
18. History of Grade 3 or higher immune mediated adverse events that were considered drug related to prior immunotherapy (e.g., checkpoint inhibitors, co stimulatory agents).
19. Known active central nervous system metastases. Participants with previously treated stable brain metastases may participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2031-02 (Estimated); Study Completion 2033-02 (Estimated)

PRIMARY OUTCOMES:
Phase 1 (Dose-Escalation): Recommended phase 2 dose of SB-4826 | 21 days
  To determine the recommended phase 2 dose of SB-4826, separately for each group. The recommended phase 2 dose will be the optimal biological dose based on consideration of safety (e.g., dose limiting toxicity, maximum tolerated dose, treatment-related adverse events) information together with all available pharmacokinetics, pharmacodynamics, and efficacy data. The recommend phase 2 dose will not exceed the maximum tolerated dose, which is the dose-level determined by the Bayesian Optimal Interval design with a target toxicity rate of 30% within the first 21 days.
Phase 2 (Dose-Expansion/ Combination Therapy): Efficacy of SB-4826 at the recommended phase 2 dose. | 6 months
  Objective response rate defined as the percentage of participants having a complete response or partial response within 6 months of the first dose of study therapy, as determined by investigator assessment per 2016 Lugano Classification criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Vu, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available.